CLINICAL TRIAL: NCT03824600
Title: Physiological Patterns of Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Jeroen Sonck, Co-Director Catheterization Laboratory, Onze Lieve Vrouw Hospital
Other Study IDs: CRI-0002
Record Dates: First submitted 2019-01-27; First posted 2019-01-31 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fractional Flow Reserve Motorized Pullback — A pullback device (Volcano R 100, San Diego CA, USA), adapted to grip the coronary pressure wire (PressureWire X, St Jude Medical, Minneapolis, USA), set at a speed of 1 mm/sec to pullback the pressure-wire until the tip of the guiding catheter during continued pressure recording.

SUMMARY:
Registry of patients undergoing invasive fractional flow reserve measurement using a motorized device.

DETAILED DESCRIPTION:
A prospective registry of patients undergoing clinically indicated coronary angiography with fractional flow reserve evaluation for vessels with intermediate coronary lesions defined as visual diameter stenosis between 30% and 70%. A motorized fractional flow reservepullback evaluation will be performed at the discretion of the operators. The objective of the present study is to describe the physiological patterns of coronary artery disease using motorized coronary pressure pullbacks during continuous hyperemia in patients with stable coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary artery disease

Exclusion Criteria:

* acute coronary syndromes
* previous coronary artery bypass grafting
* significant valvular disease
* severe obstructive pulmonary disease or asthma bronchial
* severe tortuosity or severe calcification

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing clinically indicated coronary angiography and fractional flow reserve evaluation for intermediate coronary lesions defined as visual diameter stenosis between 30% and 70%
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Physiological Patterns of Coronary Artery Disease (i.e. focal, diffuse or combined) | Immediate post-procedure. No follow-up is schedule for this trial.
  Describe the physiological patterns of coronary artery disease using motorized coronary pressure pullbacks during continuous hyperemia in patients with stable coronary artery disease. A pullback device adapted to grip the coronary pressure wire with a speed of 1 mm/sec during continued pressure recording will be used. A fractional flow reserve value every 100 microns will be extracted from the pressure tracing and plotted against the length to generate a pullback curve. Fractional flow reserve will be defined as the ratio of the moving average of the proximal and distal coronary pressures. The patterns of physiological disease will be classified as focal or diffuse according to the visual inspection of the fractional flow reserve pullback curve. The patterns of coronary artery disease will be reported as a focal, diffuse or combined pattern (i.e. focal and diffuse).

OTHER OUTCOMES:
Classification of the physiological patterns of coronary artery disease using a quantitative metric | Immediate post-procedure. No follow-up is schedule for this trial.
  Based on the data obtained using the fractional flow reserve pullbacks and conventional coronary angiography a quantitative classification of the physiological pattern of coronary artery disease based on the functional contribution of the epicardial lesion (i.e. lesion-related pressure drop) with respect to the total vessel fractional flow reserve will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard De Bruyne, MD, PhD, Study Chair — OLV-Aalst
Locations (2):
- Belgium (2):
  - OLV Aalst, Aalst, West Flanders
  - University of Brussels, Brussels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Argacha JF, Decamp J, Vandeloo B, Babin D, Lochy S, Van den Bussche K, de Hemptinne Q, Xaplanteris P, Magne J, Segers P, Cosyns B. Guiding Myocardial Revascularization by Algorithmic Interpretation of FFR Pullback Curves: A Proof of Concept Study. Front Cardiovasc Med. 2021 Mar 11;8:623841. doi: 10.3389/fcvm.2021.623841. eCollection 2021. PMID 33778020
- [Derived] Collet C, Sonck J, Vandeloo B, Mizukami T, Roosens B, Lochy S, Argacha JF, Schoors D, Colaiori I, Di Gioia G, Kodeboina M, Suzuki H, Van 't Veer M, Bartunek J, Barbato E, Cosyns B, De Bruyne B. Measurement of Hyperemic Pullback Pressure Gradients to Characterize Patterns of Coronary Atherosclerosis. J Am Coll Cardiol. 2019 Oct 8;74(14):1772-1784. doi: 10.1016/j.jacc.2019.07.072. PMID 31582137